CLINICAL TRIAL: NCT02650778
Title: Automated Breast Ultrasound Screening in Women With Dense Breasts (BIRADS 3 or 4) and BIRADS Category 1 or 2 Mammogram Assigning BIRADS 3 Lesions to Yearly Follow-up
Brief Title: Automated Breast Ultrasound Screening
Acronym: ABUS
Status: Completed | Type: Observational
Sponsor: Northeastern Ohio Radiology Research and Education Fund (Other)
Responsible Party: Principal Investigator, Richard G. Barr MD, PhD, Medical Director, Northeastern Ohio Radiology Research and Education Fund
Other Study IDs: 13-06-0007
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Automated whole breast ultrasound; BI-RADS category 3 lesions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Breast ultrasound — automated whole breast ultrasound

SUMMARY:
Women with dense breasts (BIRADS 3 or 4) with a BIRADS category 1 or 2 mammogram are asked to participate in a automated volume breast ultrasound scanner. The study evaluates prospectively the changes in recall rate, positive biopsy rate, cancer detection rate when BIRADS category 3 lesions are given a 1 year follow-up recommendation.

DETAILED DESCRIPTION:
Women with dense breasts (BIRADS 3 or 4) with a BIRADS category 1 or 2 mammogram are asked to participate in a automated volume breast ultrasound scanner. If the women agrees to participate and sign informed consent she undergoes an automated whole breast scan. The scan is interpreted independent of the mammogram. Scans are assigned a BIRADS category score of 1, 2, 3,or 0. BIRADS category 3 lesions are reported as no evidence of malignancy and a 1 year follow-up is recommended. BIRADS category 0 lesions are requested to have a hand held ultrasound including elastography. Follow up is then determined by BIRADS score and elastography results of hand held ultrasound.

The study evaluates prospectively the changes in recall rate, positive biopsy rate, cancer detection rate when BIRADS category 3 lesions are given a 1 year follow-up recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Women age >18 scheduled for routine screening mammogram. Women with Density 3 or 4 and BIRADS category 1 or mammogram are asked to participate in study

Exclusion Criteria:

* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women age >18 scheduled for routine screening mammogram. Women with Density 3 or 4 and BIRADS category 1 or mammogram are asked to participate in study
Sampling Method: Non-Probability Sample
Enrollment: 2257 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Decreased recall rate for screening breast ultrasound while maintaining cancer detection rate | 3 years

SECONDARY OUTCOMES:
Increased positive biopsy rate | 3 years

REFERENCES:
- [Derived] Barr RG, DeSivestri A, Golatta M. Outcomes of Return to Routine Screening for BI-RADS 3 Lesions Detected at Supplemental Automated Whole-Breast Ultrasound in Women With Dense Breasts: A Prospective Study. AJR Am J Roentgenol. 2021 Dec;217(6):1313-1321. doi: 10.2214/AJR.21.26180. Epub 2021 Jul 14. PMID 34259039